CLINICAL TRIAL: NCT04316299
Title: Acute Kidney Injury in Patients Hospitalized With COVID-19 in Wuhan, China: a Single-center Retrospective Observational Study
Brief Title: Acute Kidney Injury in Patients Hospitalized With COVID-19
Status: Completed | Type: Observational
Sponsor: Zhenhua Zen (Other)
Responsible Party: Sponsor-Investigator, Zhenhua Zen, Associate Professor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Other Study IDs: hkyy2020-005 AKI
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: COVID-19; Acute Kidney Injury; Kidney Function
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI: COVID-19 patients with acute kidney injury
- non-AKI: COVID-19 patients without acute kidney injury

SUMMARY:
The kidney may be affected in coronavirus-2019 disease (COVID-19). This study assessed the predictors and outcomes of acute kidney injury (AKI) among individuals with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 pneumonia patients diagnosed by WHO criteria

Exclusion Criteria:

* Patients who were younger than 18 years,
* Patients who had undergone renal replacement therapy (RRT) before admission,
* Patients whose entire stay lasted for less than 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Hankou Hospital in Wuhan with confirmed COVID-19 pneumonia from 5th Jan to 28th Feb.
Sampling Method: Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-08 (Actual)

PRIMARY OUTCOMES:
Rate of Acute Kidney Injury | From date of admission until the date of discharge or death from any cause, up to 60 days
  the incidence of Acute Kidney Injury

SECONDARY OUTCOMES:
Rate of Death | From date of admission until the date of death from any cause, up to 60 days
  death from any cause in the hospital
the length of hospital stay | From date of admission until the date of discharge or death from any cause, up to 60 days
  days from admission to discharge or death

CONTACTS AND LOCATIONS:
Locations (1):
- Hankou Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided